CLINICAL TRIAL: NCT06149585
Title: Changes in Microbial Status From Dentate, Edentulous and After Dental Implant Placement
Status: Recruiting | Type: Observational
Sponsor: Case Western Reserve University (Other)
Responsible Party: Sponsor
Other Study IDs: STUDY20221051
Record Dates: First submitted 2023-11-13; First posted 2023-11-29 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-06

CONDITIONS: Edentulous Mouth; Periodontal Diseases; Periodontitis, Adult; Microbial Colonization
MeSH Terms: conditions — Mouth, Edentulous; Periodontal Diseases; Chronic Periodontitis; Communicable Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Separate pooled samples will be collected from 3 areas of the mouth: oral mucosa, tongue, Peri-implant sulci (when applicable). Surfaces will be swabbed for 30 seconds each with a single CatchAll™ Swab. Care will be taken to avoid contacting the teeth. The swab will be immediately swirled in 400 uL Tris-EDTA buffer, pressing the swab against the tube walls for 20 seconds to transfer the material to the solution. The swab will be then discarded. The procedure will be repeated, but this time swabs will be placed in 400 uL of RNA Cell Protect (Qiagen). Subgingival plaque collection: The subgingival plaque will be then sampled with a Gracey curette obtaining samples from all available surfaces, and placed in 400 uL of TE buffer or 400 uL RNA Cell Protect (Qiagen). Samples will be immediately transferred to a -80 degree C freezer until further processed.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Intra-Lock Fusion Implants: These patients will receive Intra-Lock Fusion Implants during implant placement
  Interventions: Other: Microbial Sampling
- Tapered Pro Implants: These patients will receive Tapered Pro Implants during implant placement
  Interventions: Other: Microbial Sampling

INTERVENTIONS:
Other: Microbial Sampling — Pool microbial sampling will be performed and changes in the microbiome will be evaluated and compared for differences

SUMMARY:
The objectives of this study are to analyze the oral microbiome modulations occurring during the transition from partial (with some residual teeth) to full edentulous (without remaining teeth) status and implant placement in subjects affected by severe periodontitis; to evaluate if microbiome changes in relation to the used of different implant material/surface; and to assess the variance of the changes to determine the sample size for future longitudinal prospective studies.

DETAILED DESCRIPTION:
The introduction of dental implants has significantly changed the treatment approach for prosthetic rehabilitation of partially and edentulous patients. In the last decades an increasing number of patients have received implants for the replacement of missing teeth. Although dental implants have proved to be a very predictable treatment option, in the long term they are susceptible to biologic complications that may lead to implant loss. In particular, two major peri-implants conditions have been described: peri-implant mucositis and peri-implantitis. Peri-implant mucositis is an inflammatory condition of the peri-implant tissue without bone loss and is considered reversible once the biofilm is removed; Peri-implantitis is an inflammatory condition that affect the bone support of the implant and if untreated may lead to implant loss. The major etiologic factors involved in Peri-implantitis are: history of periodontitis, poor plaque control, and poor patient compliance. The high susceptibility to biologic complication of implants placed in partially edentulous patients with history of periodontitis has been demonstrated in several studies. Multiple studies demonstrated periodontal pathogens can transfer from teeth to implants. However, it is unclear whether the same occurs on implants placed in edentulous subjects that have lost their dentition due to periodontitis. Previous investigations have shown a significant reduction but not the complete elimination of putative periodontal pathogens following full mouth extractions. Most of the studies on microbial population around teeth and implants are based on assessing the presence or absence of putative pathogens. Limited information is available regarding the whole microbiome shift from dentate to edentulous status and the changes occurring around the implant crevice after implants are placed. The use of 16S RNA pyrosequencing has been recently introduced to study the oral microbiome in health and disease. More recently shotgun metagenomic sequencing was introduced which allows evaluation of all the genes in a microbial community thereby revealing information on community composition and also community functional capacity. Shotgun sequencing also allows tracking of strains using single nucleotide variants or gene-content assessments, allowing assessment of longitudinal changes in colonization. The purpose of this investigation is to assess the oral microbiome changes in subjects with terminal dentition due to periodontitis over the entire treatment period, including the shift from dentate status to edentulous and finally post-implant.

Patients diagnosed with terminal dentition due to periodontitis with the intention to replace the dentition with implant-supported/retained restorations will be invited to participate.

Visit 1 - Screening visit to evaluate patient qualification for the study. Inclusion-Exclusion criteria. Qualifying patients will be enrolled and will receive a full mouth examination including an assessment of PD, clinical attachment level (CAL), BoP, and furcation involvement.

Visit 2 - Baseline microbial sampling and Full mouth extractions. Pool microbial sampling will be performed before teeth extractions. An immediate denture may be delivered at this time.

Visit 3 - Diagnostics for Implant Placement 3-4 months after teeth extraction. Diagnostic appointments may include multiple visits for diagnostics setup, Cone-beam computed tomography (CBCT), and provisional denture adjustments prior to implant placement.

Visit 4 - Mucosal-oral microbial sampling Implant Placement. Pool microbial sampling will be performed immediately before implant placement. Intra-Lock Fusion Implants or Tapered Pro Implants (Bio Horizon) will be alternatively allocated to each participant. Implants will be submerged for a 2 stage of healing. A Standard peri-apical X-ray of the implants will be taken.

Visit 5 - follow-up after implant placement and suture removal this will take place 14 days after implant placement.

Visit 6 - Implant uncover. 3-4 months after implant placement abutments will be connected to the implants after a 2nd stage uncover surgery Visit 7 - follow up after implant uncover and suture removal will take place 14 days after implant uncover procedure.

Visit 8 - Restorative connection *. The permanent abutments will be connected to the implants, at this stage, a pooled microbial sample will be collected. Baseline implant probing depth (PD), keratinized mucosa (KM), and bleeding on probing (BoP) will be recorded. Standardized peri-apical X-ray of the implants will be taken. Visit 9 - 6 Months post-loading, Pooled Microbial sampling, PD, KM, and BoP will be recorded, Standardized periapical X-ray of the implants Visit 10 - 12 Months post-loading, Pooled Microbial sampling, PD, KM and BoP will be recorded. Standardized peri-apical X-ray of the implants will be taken.

Pooled Microbial samples: At visits 2, 4,8,9,10. Separate pooled samples will be collected from 3 areas of the mouth: oral mucosa: swabs from oral mucosa including upper and lower lips and left and right buccal surfaces tongue: swab from tongue dorsum Peri-implant sulci (when applicable), plaque collection using curettes around implants Swab from oral mucosa and tongue: Oral mucosa and tongue will be swabbed using a separate sterile sponge swab. Surfaces will be swabbed for 30 seconds each with a single CatchAll™ Swab. Care will be taken to avoid contacting the teeth. The swab will be immediately swirled in 400 uL Tris-EDTA buffer, pressing the swab against the tube walls for 20 seconds to transfer the material to the solution. The swab will be then discarded. The procedure will be repeated, but this time swabs will be placed in 400 uL of RNA Cell Protect (Qiagen). Samples will be immediately transferred to a -80C freezer until further processed. Subgingival plaque collection: Prior to the collection of subgingival plaque at a tooth or implant site, supragingival plaque will be removed with a Gracey curette. The subgingival plaque will be then sampled with a new Gracey curette obtaining samples from all available surfaces, and placed in 400 uL of Tris-Ethylenediaminetetraacetic acid (EDTA) (TE) buffer or 400 uL RNA Cell Protect (Qiagen). Samples will be immediately transferred to a -80C freezer until further processed. 4. Medical and dental history form from Axium. 5. Single CatchAll™ is a sterile cotton tip applicator. The periodontal curette is a type of hand-activated instrument used in dentistry and dental hygiene for the purpose of scaling and root planing. The periodontal curette is considered a treatment instrument. Periodontal curettes have one face, one or two cutting edges and a rounded back and rounded toe.

Only the microbial sampling is being done for research purposes. The other procedures described above are standard of care and the subjects would receive it even if they were not in the study

ELIGIBILITY:
Inclusion Criteria:

1. At least 21 years of age
2. Diagnosis of Stage III or IV periodontitis based on full mouth probing and full mouth x-rays
3. Planned for full mouth extraction and replacement by dental implants.
4. Rehabilitation with Implant supported restorations either maxilla and/ or mandible.
5. At least 2 implants available for examination.
6. No bone augmentation required.

Exclusion Criteria:

1. Conditions requiring chronic routine prophylactic use of antibiotics.
2. Conditions requiring prolonged use of steroids.
3. History of leukocyte dysfunction and deficiencies
4. Bleeding disorders
5. History of neoplastic disease requiring use of radiation or chemotherapy
6. Metabolic bone disorders
7. Uncontrolled endocrine disorder
8. Use of any investigational drug or device within the 30 day period prior to implant surgery.

10. Alcoholism or drug abuse 11. Patient infected with HIV 12. Condition or circumstances, in the opinion of the investigator, which would prevent completion of study participation or interfere with analysis of study results, such as history of non-compliance, unreliability.

Local Exclusion Criteria

1. Local inflammation
2. Mucosal disease such as erosive lichen planus
3. History of local irradiation therapy
4. Osseous lesion.
5. Active infection with suppuration or fistula track.
6. Persistent intraoral infection different than periodontitis

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population will consist of patients with stage III or IV periodontitis who are patients at the Case Western Reserve University School of Dental Medicine in the Department of periodontitis who are seeking to remove all of their remaining teeth and replace the teeth lose to periodontal disease with dental implants
Sampling Method: Non-Probability Sample
Enrollment: 12 (Estimated)
Dates: Start 2023-08-16 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2027-05-01 (Estimated)

PRIMARY OUTCOMES:
Oral microbiome composition changes in patients who are dentate, edentulous, and have dental implants | Through study completion, an average of 24 months
  To analyze the oral microbiome modulations through DNA analysis of microbial samples occurring during the transition from partial (with some residual teeth) to full edentulous (without remaining teeth) status and implant placement in subjects affected by severe periodontitis
Oral microbiome changes in two different implant platform types | Through study completion, an average of 24 months
  To evaluate if microbiome changes through DNA analysis of microbial samples in relation to the use of different implant material/surface

SECONDARY OUTCOMES:
Sample size | Through study completion, an average of 24 months
  To assess the variance of the changes to determine the sample size for future longitudinal prospective studies

CONTACTS AND LOCATIONS:
Overall Officials: Gian Pietro Schincaglia, DDS,PhD, Principal Investigator — Case Western Reserve University
Locations (1):
- Case Western Reserve University Department of Periodontics, Cleveland, Ohio, United States